CLINICAL TRIAL: NCT00249327
Title: Online HIV Prevention Vignette Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Solutions (Other)
Collaborators: Van Ameringen Foundation Inc (Other); The New York Community Trust (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 063005
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: HIV Infections
Keywords: HIV testing; HIV disclosure; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Educational Status

INTERVENTIONS:
Behavioral: education

SUMMARY:
This is an evaluation of the effect that an online live action, dramatic vignette about four gay men, two HIV positive and two HIV negative, struggling with the responsibility for safer sex has on the sexual behavior and HIV testing intentions of the gay/bisexual men who watch the vignette and participate in the evaluation study. The primary hypothesis is that men will be more likely to: 1)express the intent to have an HIV test and 2) to express the intent to inform their sex partners of their HIV status after watching the vignette. The secondary hypothesis is that men will be more likely to follow through on these intentions in the three months following the intervention than they were in the three months before viewing the vignette. This is a one group pre-posttest intervention in which each man serves as his own control.

DETAILED DESCRIPTION:
* Men over 18 years of age will be recruited for the study through a banner posted on the exit page of manhunt.net an internet gay hook-up site. Those clicking on the banner will go to the evaluation website (www.hivbigdeal.org)
* asked to read the consent and click agreement.
* asked to complete a relatively brief questionnaire about their sexual behavior, HIV testing and HIV disclosure in the preceding three months
* watch the 8 minute dramatic vignette
* complete a brief questionnaire that elicits their response to the video and their HIV testing and disclosure intentions.
* if they agree to provide the study with their e-mail address, participants will be re-contacted in three months and asked to complete a second behavioral survey online that asks about sexual behavior, HIV testing and HIV disclosure in the three months since watching the vignette.Behavior before and after watching the vignette will be compared.
* The entire study will be conducted online.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Gay/bisexual men
* Age > 18

Exclusion Criteria:

* Women
* Men under 18
* Men who do not have sex with other men

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2005-10; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Increase in HIV testing
Increase in disclosure of HIV status to sex partner

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Chiasson, DrPH, Principal Investigator — Medical and Health Research Association of New York City Inc.
Locations (1):
- Medical and Health Research Association of New York City, Inc., New York, New York, United States